CLINICAL TRIAL: NCT02738788
Title: Assessing Intraoperative Airway Changes and Their Regression to Baseline in Patients Undergoing Elective Surgical Procedures in the Prone and Trendelenburg Positions
Brief Title: Airway Changes in Patients Undergoing Elective Surgical Procedures in the Prone and Trendelenburg Positions
Status: Active, not recruiting | Type: Observational
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 11705
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Airway Management
Keywords: airway; airway changes; MMS; prone position; Trendelenburg position
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Intubation — The patient's airway will be visually assessed and photographed while the patient is resting comfortable in bed with the head up at 30-45 degrees and classified into one of 4 MMS categories. Digital photographs will be taken and the stored image prepared by the investigators in such a way that the patient cannot be individually identified (mouth only).
  Neck circumference will be measured at the level of the thyroid cartilage using a tape measure, with temporary ink marks on the skin to allow for subsequent measurements at the same point.
  After the patient has been extubated and recovered in the PACU for 30 minutes, their airway will be re-assessed and documented. These evaluations will be repeated at 2, 3, and 4 hours, as well as the next morning.

SUMMARY:
The goal of this study is to track the intraoperative changes that occur in the airways of patients undergoing 1) laparoscopic surgeries in the Trendelenburg position, and 2) spinal surgeries in the prone position, as well as the regression of these changes postoperatively. These surgeries are known to cause edema and swelling of the soft tissues of the head and neck, temporarily worsening airway anatomy, but there is little data quantifying these changes, and no studies have investigated the time course required for the airway to return to its baseline after extubation. This would be important clinical information given that airway management is always a major concern perioperatively. The investigators will test hypotheses by evaluating patients' airways preoperatively, immediately post-extubation, and at regular intervals thereafter using the Modified Mallampati Score class (MMS), in which a patient's airway is scored from class 1 to 4 (in which 4 indicates the highest likelihood of a difficult intubation) based on the visibility of the soft palate, uvula, and faucial pillars inside the oral cavity.

DETAILED DESCRIPTION:
Background: One of the primary methods to assess airway dimension changes is the Modified Mallampati Score (MMS). MMS has been a valuable tool in assessing difficulty of intubation in previous studies as it is a simple, reproducible, and reliable preoperative and preanesthetic assessment of oral volume. MMS is evaluated by asking the patient to open their mouth and protrude their tongue without phonation. A score on a scale of 1-4 is assigned based on identifiable intraoral anatomic structures. MMS scores of 3 and 4 are strongly associated with difficult laryngoscopy and intubation.

Extensive observational research in the obstetric population has demonstrated that airway changes, including increasing MMS and decreasing oropharyngeal volume, occur during labor. It has been found that 63% of parturients experienced an increase in MMS over the course of their labor, with the fraction of patients scoring 3 or 4 peaking at 51.7%, compared with only 10.3% early in labor. Notably, of those patients that reached a class 4, 21% remained at that classification 48 hours postpartum. It has been found that 18% of patients whose airway class worsened during labor had not returned to their prelabor class 36-48 hours after delivery.

These obstetric findings have prompted a limited number of studies investigating airway changes in patients undergoing surgical procedures. This study will focus on surgeries in the prone and Trendelenburg positions, as they would intuitively predispose patients to edema and fluid retention in the head and neck. MMS increased in 78% of patients, with 29% increasing by two or more classes in patients undergoing lumbar spine surgery in the prone position. Furthermore, although laparoscopic surgery has been shown to increase lung and chest wall mechanical impedance, which leads to increases in abdominal and intrathoracic pressure, as well as an increase in central venous pressure with subsequent increases in intraocular pressure, no studies have been performed to specifically track resultant airway changes. Lastly, to investigators' knowledge no studies have investigated the postoperative resolution of airway changes after either type of procedure.

Rationale: There is evidence, both investigational and anecdotal, that airway changes may occur during certain surgeries or procedures, and that patient positioning may play a large role in precipitating them. However, research on this phenomenon in the surgical population, unlike the obstetric population, is sparse. Similarly, investigations into the time required for airway changes to regress back to baseline has been included in a number of obstetric airway studies, but not in any surgical ones. Lastly, it has been suggested that other surgical factors, such as fluid balance or procedure duration, may alter the degree of airway changes, but results from the few recent studies on the topic have been unclear. Thus, this study seeks to further investigate the influence of prone and Trendelenburg positioning, as well as surgical variables, on perioperative airway changes, and quantify the time required for patients' airways to return to their preoperative state.

Based on clinical observation, the primary hypothesis is that there will be a significant difference between mean scoring class change between 2 study groups from preoperative baseline to initial postoperative assessment. Investigators hypothesize that T-burg surgery patients will have a mean change of 2 classes compared to a mean change of only one class for prone spine surgery patients.

The secondary hypothesis is that airway changes occurring in patients undergoing prone procedures will resolve significantly sooner than (3 - 4 hours) than those of patients undergoing Trendelenburg surgeries (> 4 hours).

Thirdly investigators will investigate the effects of demographic, physiological, and surgical & anesthetic variables on postoperative MMS changes and their resolution.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for elective spinal surgery in the prone position or laparoscopic or surgery in the Trendelenburg position.

Exclusion Criteria:

* Patients with a preoperative MMS of 4, existing oropharyngeal pathology, or the inability to fully open their mouth, or severely limited neck mobility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over the age of 18 undergoing scheduled spinal surgery in the prone position or laparoscopic or surgery in the Trendelenburg position.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in MMS after surgery | 1-4 hours after surgery
  Based on institutional observations, we expect both prone and Trendelenburg patients to exhibit significant airway changes/increases in MMS after surgery. Additionally, we expect to find that these changes will require approximately 4 hours to fully regress, and that perioperative and intraoperative factors, such as IV fluid and steroid administration, will affect both the degree of airway changes and the time course of their regression.

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No